CLINICAL TRIAL: NCT05535036
Title: Intravenous Dexamethasone: Postoperative Analgesic Effect in Caesarean Section Under Spinal Anesthesia
Brief Title: Intravenous Dexamethasone Effectiveness in Post Caesarean Section Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, clinical Professor, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: dexa C section
Record Dates: First submitted 2022-08-30; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Cesarean Section; Dexamethasone; Postoperative Pain; Spinal Anesthesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexamethasone group (Experimental): patients received 8mg(2ml) of intravenous dexamethasone after spinal anesthesia
  Interventions: Drug: Dexamethasone 4mg
- placebo group (Placebo Comparator): patients received 2ml of a saline solution after spinal anesthesia
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone 4mg — all patients had standard non-invasive monitoring including an electrocardiogram, non invasive blood pressure and pulse oxymetry. An 18-gauge intravenous cannula was inserted into the nondominant arm or hand and 500 ml of a saline solution (0.9 %) was infused. The prevention of postoperative nausea and vomiting (PONV) was assured to all patients by administering 4 mg of IV Ondansetron. Spinal anesthesia was performed according to our department protocol: L4-L5 or L3-L4 intervertebral space puncture using a 25 gauges needle, with injection of 0.5% hyperbaric Bupivacaine mixture (dose depending on patient height) associated with 2.5 ug Sufentanil and 100 ug Morphine. Before surgical incision, patients received either an intravenous injection of 8 mg (2 ml) Dexamethasone (DG) or 2 ml of a Saline solution (PG).
  Arms: dexamethasone group
Drug: Placebo — patients received 2ml of intravenous saline solution
  Arms: placebo group

SUMMARY:
The management of postpartum pain is essential to ensure early rehabilitation for parturients. Intravenous dexamethasone has a potent analgesic action when used in the context of general anesthesia. Nevertheless, it remains poorly studied in combination with spinal anesthesia (SA). The aim of this study was to assess the analgesic effect of intravenous dexamethasone after caesarean section under SA.

Methods: We conducted a prospective, randomized, double-blinded study including 84 ASA II-III parturient at term who were proposed for caesarean section under SA. Parturient were randomized into two groups: Dexamethasone group (DG) who received 8mg of intravenous dexamethasone (2ml) immediately after SA and placebo group (PG) who received 2ml of isotonic saline. The analgesic protocol was standardized and we opted for Tramadol as rescue analgesic. The main outcome is the use of Tramadol in the first 24 hours postpartum..

DETAILED DESCRIPTION:
A a prospective randomized double-blinded controlled study including 84 parturient women, conducted at the Anesthesia and Surgical Intensive Care Department of Mongi Slim University Hospital, La Marsa Tunisia. It was performed after obtaining the approval of the Research Ethical Committee of our hospital (Ethical Committee No. 02/2020). Eligible patients were informed of the study design and their written consent was obtained.

Patients:

Inclusion criteria were Age >= 18 years, American Society of Anesthesiologists (ASA) statue II-III, a pregnancy term >= 37 weeks, elective cesarean section and Pfannenstiel incision.

Exclusion criteria were severe hypertension / preeclampsia, poorly balanced diabetes mellitus, allergy to one of the study drugs, patients with chronic pain or long-term use of opioids, and patients on long-term corticosteroid therapy.

Study protocol During the preoperative visit, all patients have had a full clinical examination and further examinations have been requested in accordance with the most recent guidelines. The informed written consent was obtained at this moment. Postoperative pain predisposition (the prediction of pain and the anxiety level) was assessed using a questionnaire.

Randomization and allocation were performed using a computer-generated sequence of randomization numbers and the envelope technique; patients were randomized into two groups:

* Dexamethasone Group (DG): receiving 8mg (2ml) of intravenous (IV) Dexamethasone after spinal anesthesia
* Placebo Group (PG): receiving 2 ml of IV Saline solution after spinal anesthesia.

Patients enrolled and the anesthesiologists in charge were both blinded to the study group. In the operating room, all patients had standard non-invasive monitoring including an electrocardiogram, non invasive blood pressure and pulse oxymetry. An 18-gauge intravenous cannula was inserted into the nondominant arm or hand and 500 ml of a saline solution (0.9 %) was infused. The prevention of postoperative nausea and vomiting (PONV) was assured to all patients by administering 4 mg of IV Ondansetron. Spinal anesthesia was performed according to our department protocol: L4-L5 or L3-L4 intervertebral space puncture using a 25 gauges needle, with injection of 0.5% hyperbaric Bupivacaine mixture (dose depending on patient height) associated with 2.5 ug Sufentanil and 100 ug Morphine. Before surgical incision, patients received either an intravenous injection of 8 mg (2 ml) Dexamethasone (DG) or 2 ml of a Saline solution (PG). During the procedure, we noted hemodynamic constants, surgical related data and APGAR score for the newborns. At the end, patients were transferred initially to the post-operative monitoring room, and then to the Gynecology Obstetric department after assessing the hemodynamic constants, the absence of bleeding, the good tone of the uterine globe and the disappearance of the motor block.

The analgesic protocol was standardized: systemic analgesia during the first 24 hours was assured by a postoperative regimen combining intravenous Paracetamol 1g*4/day and Nefopam 20 mg*3/day . The rescue analgesic is IV Tramadol 100 mg administered at the request of the patient and if the analog visual scale (AVS) was greater than 3/10, with a maximum dose of 100 mg * 3/day. Static and dynamic pain was assessed at 2 hours, 6 hours, 12 hours and 24 hours postoperatively using the analog visual scale ( values raging from 0 for no pain to 10 for a maximum pain). Time to first request and cumulative dose of Tramadol were recorded. We also noted the length of the sensory and the motor blocks, postoperative nausea and vomiting and patient satisfaction. Hospital discharge was allowed after 24 hours if there were no complications.

Follow-up at 3 months:

Patients were contacted after 3 months to complete a telephonic survey about chronic pain and postpartum depression . We excluded patients who had other surgery within 3 months of the cesarean section or any other cause of chronic pain.

Outcomes:

Our main outcome was the use of Tramadol within the first 24 hours. Secondary endpoints were static and dynamic analog visual scale at 2 hours, 6 hours,12 hours, and 24 hours, time to first request of Tramadol, cumulative Tramadol dose within the first 24 hours, length of sensory and motor block, incidence of post-operative nausea and vomiting (PONV), chronic pain at 3 months, incidence of postpartum depression, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) statue II-III,
* a pregnancy term >= 37 weeks
* elective cesarean section
* Pfannenstiel incision

Exclusion Criteria:

* severe hypertension / preeclampsia
* poorly balanced diabetes mellitus
* allergy to one of the study drugs
* patients with chronic pain or long-term use of opioids
* patients on long-term corticosteroid therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
tramadol requirements | 24 hours
  The rescue analgesic was IV Tramadol 100 mg administered at the request of the patient and if the analog visual scale (AVS) was greater than 3/10, with a maximum dose of 100 mg * 3/day.

SECONDARY OUTCOMES:
pain scores | H2, H6, H12 and H24
  Static and dynamic pain was assessed at H2, H6, H12, and H24 postoperatively using the AVS ( analog visual scale)
postoperative nausea and vomiting(PONV) | 24 hours
  we assessed the occurence of postoperative nausea and vomiting during the first 24 hours after surgery
Chronic pain | 3 months
  we performed a telephonic questionnaire to assess chronic pain

CONTACTS AND LOCATIONS:
Locations (1):
- Mongi Slim University Hospital, La Marsa, Tunis Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: No